CLINICAL TRIAL: NCT01922258
Title: A Phase 3, 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Flexible Dosing of Brexpiprazole (OPC-34712) in the Treatment of Subjects With Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: Safety and Tolerability Study of Flexible Dosing of Brexpiprazole in the Treatment of Subjects With Agitation Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-12-284
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Agitation Associated With; Alzheimer's Disease; Alzheimer's Type; Mental Disorder; Nervous System Diseases
Keywords: OPC-34712; brexpiprazole; Dementia; Alzheimer's Disease; Cognitive Disorders; Agitation
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders; Nervous System Diseases; Dementia; Cognitive Dysfunction; Psychomotor Agitation | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo Once-Daily
  Interventions: Drug: Brexpiprazole, OPC-34712
- Brexpiprazole (flexible dose range 0.5 to 2 mg) (Experimental): Titrate up from 0.25 mg/day brexpiprazole to 1 mg/day brexpiprazole. After achieving 1 mg/day target dose may be increased or decreased based on efficacy and tolerability. Allowable flexible doses will be 0.5 mg/day, 1 mg/day, or 2 mg/day.
  Interventions: Drug: Brexpiprazole, OPC-34712

INTERVENTIONS:
Drug: Brexpiprazole, OPC-34712 — Flexible dose of 0.5 to 2 mg/day or placebo tablets for up to 12 weeks

SUMMARY:
To compare the efficacy of flexible dosing of brexpiprazole with placebo in subjects with agitation associated with dementia of the Alzheimer's type

DETAILED DESCRIPTION:
Behavioral symptoms, such as agitation, are core features in subjects with Alzheimer's disease and related dementias and develop in the majority of dementia subjects. The presence of agitation in subjects with Alzheimer's disease places a significant burden not only on subjects and their caregivers but also on the healthcare system.

This is a trial designed to assess the safety and efficacy of flexible dosing of brexpiprazole in the treatment of subjects with agitation associated with dementia of the Alzheimer's type. The trial consists of a 12-week double-blind treatment period with a 30-day follow-up. The trial population will include male and female subjects between 55 and 90 years of age (inclusive) with a diagnosis of probable Alzheimer's disease, who are residing either in an institutionalized setting or in a non-institutionalized setting where the subject is not living alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 55 to 90 years of age, inclusive, at the time of informed consent.
* Subjects who are residing at their current location for at least 14 days before screening and are expected to remain at the same location for the duration of the trial.
* Subjects with diagnosis of probable Alzheimer's disease according to NINCDS-ADRDA criteria.
* Subjects with a MMSE score of 5 to 22, inclusive, at screening and baseline visits.
* Subjects with onset of symptoms of agitation at least 2 weeks prior to the screening visit.
* Subjects with a total score greater than or equal to 4 on the agitation aggression item of the NPI-NH or NPI/NPI-NH at the screening and baseline visits.
* Subjects who require pharmacotherapy for the treatment of agitation per the investigator's judgement, after an evaluation of reversible factors (eg, pain, infection, polypharmacy) and a trial of nonpharmacological interventions.
* Subjects must have a previous MRI or CT scan of the brain, which was performed after the onset of symptoms of dementia, with findings consistent with the diagnosis of Alzheimer's disease.

Exclusion Criteria:

* Subjects with dementia or other memory impairment not due to Alzheimer's disease.
* Subjects with history of stroke, well-documented transient ischemic attack, or pulmonary or cerebral embolism.
* Subjects who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, gastrointestinal, or psychiatric disorders.
* Subjects who have been diagnosed with an Axis I disorder (DSM-IV-TR criteria).
* Subjects with uncontrolled hypertension.
* Subjects with uncontrolled insulin-dependent diabetes mellitus (IDDM)
* Subjects with epilepsy or a history of seizures.
* Subjects considered in poor general health based on the investigator's judgment.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Koheygi, MD, Study Director — Otsuka Pharmaceutical Development and Commercialization, Inc.
Locations (60):
- United States (24):
  - Imperial, California
  - Lakewood, California
  - Long Beach, California
  - Panorama City, California
  - Universal City, California
  - Denver, Colorado
  - Bradenton, Florida
  - Miami, Florida
  - Orange City, Florida
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Honolulu, Hawaii
  - Indianapolis, Indiana
  - Quincy, Massachusetts
  - South Dartmouth, Massachusetts
  - Ann Arbor, Michigan
  - Brooklyn, New York
  - Buffalo, New York
  - New Hyde Park, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Austin, Texas
  - Dallas, Texas
  - Woodstock, Vermont
- Bulgaria (7):
  - Burgas
  - Kardzhali
  - Pazardzhik
  - Rousse
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (2):
  - Penticton, British Columbia
  - Kentville
- Finland (2):
  - Kuopio
  - Turku
- France (6):
  - Bourg-en-Bresse
  - Douai
  - Élancourt
  - Limoges
  - Nice
  - Toulouse
- Russia (4):
  - Tonnel’nyy, Stavropol Kray
  - Saint Petersburg
  - Saratov
  - Yekaterinburg
- Slovenia (3):
  - Ljubljana
  - Maribor
  - Šempeter pri Gorici
- Ukraine (8):
  - Donetsk
  - Kharkiv
  - Kherson
  - Kiev
  - Lviv
  - Poltava
  - Simferopol
  - Vinnytsia
- United Kingdom (4):
  - Crewe
  - Manchester
  - Margate
  - Torpoint

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Cummings JL, Chumki SR, Chang D, Zhang Z, Brubaker M, Hefting N, Such P, Wang D, Grossberg GT. Efficacy of Brexpiprazole in Participants with Agitation Associated with Dementia Due to Alzheimer's Disease: Pooled Analysis of Randomized Controlled Trials. Clin Drug Investig. 2026 Jan 27. doi: 10.1007/s40261-025-01517-9. Online ahead of print. PMID 41591746
- [Derived] Shah A, Kalu U, Chen D, Slomkowski M, Hobart M, Such P, Grossberg GT. Brexpiprazole side-effect profile in people with agitation in Alzheimer's dementia: a plain language summary. Curr Med Res Opin. 2026 Jan 14:1-3. doi: 10.1080/03007995.2025.2608578. Online ahead of print. PMID 41533472
- [Derived] Shah A, Estilo A, Sheridan PL, Kalu U, Chen D, Chang D, Slomkowski M, Lee D, Hefting N, Hobart M, Behl S, Such P, Brubaker M, Grossberg GT. Safety and Tolerability of Brexpiprazole in Participants with Agitation Associated with Dementia due to Alzheimer's Disease: Pooled Analysis of Three Randomized Trials and an Extension Trial. CNS Drugs. 2025 Oct;39(10):1011-1023. doi: 10.1007/s40263-025-01200-9. Epub 2025 Jul 19. PMID 40681915
- [Derived] Meunier J, Creel K, Loubert A, Larsen KG, Aggarwal J, Hefting N, Oberdhan D. Defining a clinically meaningful within-patient change threshold for the Cohen-Mansfield Agitation Inventory in Alzheimer's dementia. Front Neurol. 2024 Jul 23;15:1379062. doi: 10.3389/fneur.2024.1379062. eCollection 2024. PMID 39108660
- [Derived] Grossberg GT, Kohegyi E, Mergel V, Josiassen MK, Meulien D, Hobart M, Slomkowski M, Baker RA, McQuade RD, Cummings JL. Efficacy and Safety of Brexpiprazole for the Treatment of Agitation in Alzheimer's Dementia: Two 12-Week, Randomized, Double-Blind, Placebo-Controlled Trials. Am J Geriatr Psychiatry. 2020 Apr;28(4):383-400. doi: 10.1016/j.jagp.2019.09.009. Epub 2019 Oct 1. PMID 31708380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 62 sites in 9 countries: Bulgaria, Canada, Finland, France, Russia, Slovenia, Ukraine, the United Kingdom (UK), and the United States (US) and 270 participants were randomized. The date of the first ICF signed by a participant in this trial was 28 October 2013 and the date of the last trial observation was 30 March 2017.
Pre-assignment Details: The screening period ranged from 2 to 42 days (with an option to extend with approval of the medical monitor). The screening period was to determine the participant's eligibility and to washout prohibited concomitant pharmacotherapy prior to randomization.
Groups:
- Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day): Titrate up from 0.25 mg/day brexpiprazole to 1 mg/day brexpiprazole. After achieving 1 mg/day target, dose may be increased or decreased based on efficacy and tolerability. Allowable flexible doses will be 0.5 mg/day, 1 mg/day, or 2 mg/day.
- Placebo (Flexible Dose Range 0.5 to 2 mg/Day): Titrate up from 0.25 mg/day placebo to 1 mg/day placebo. After achieving 1 mg/day target, dose may be increased or decreased based on efficacy and tolerability. Allowable flexible doses will be 0.5 mg/day, 1 mg/day, or 2 mg/day.
Period: Overall Study
Arm/Group | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day)
Started | 133 | 137
Completed | 117 | 121
Not Completed | 16 | 16
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 9 | 2
Not completed — Met Withdrawal Criteria | 0 | 4
Not completed — Withdrawn by the Investigator | 1 | 4
Not completed — Withdrawal by participant | 5 | 5

BASELINE CHARACTERISTICS:
Population: All participants who were randomized into this trial. Participants were considered randomized when they were assigned a treatment number by interactive voice response system (IVRS) at the end of screening period. A participant who received trial treatment outside of the IVRS was not considered randomized, but safety was reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day) | Total
Number analyzed (Participants) | 133 | 137 | 270
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 24 | 19 | 43
  >=65 <75 years | 46 | 49 | 95
  >=75 years | 63 | 69 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 88 | 170
  Male | 51 | 49 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 128 | 129 | 257
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12/Early Termination in the Cohen-Mansfield Agitation Inventory (CMAI) Total Score
Description: The CMAI is widely used in clinical research for evaluation of agitation associated with Alzheimer's dementia, with reliability and validity in both institutionalized and noninstitutionalized participants. It consists of 29 items, all rated on a 1 to 7 scale (1=Never and 7=Several times in an hour), with 1 being the "best" rating and 7 being the "worst" rating. The total score is the sum of ratings for all 29 items. The possible total scores range from 29 to 203. The total score will be unevaluable if less than 24 of the 29 items are recorded. If 24 to 28 of the 29 items are recorded, the total score will be the mean of the recorded items multiplied by 29 and rounded to the first decimal place. The mean change from baseline (Day 0) to week 12 in the CMAI total score is reported. Statistical comparison of interest was brexpiprazole flexible dose versus placebo, analyzed using a mixed-effect model repeated measure approach. A decrease in score indicates improvement in symptoms.
Time Frame: From screening to week 12/early termination
Population: The intent-to-treat (ITT) population consisted of all participants in the randomized sample, who took at least 1 dose of the investigational medicinal product (IMP) and had a baseline and at least one postbaseline evaluation for the CMAI total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day)
Number analyzed (Participants) | 131 | 135
units on a scale | -18.9 (1.17) | -16.5 (1.13)
Statistical Analysis 1: Comparison: Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) vs Placebo (Flexible Dose Range 0.5 to 2 mg/Day); Test type: Superiority; p = 0.1454, Mixed-effect model repeated measure; Treatment Difference = -2.34, 95% CI 2-sided [-5.49 to 0.82]

2. Secondary Outcome: Change in the Clinical Global Impression Severity of Illness (CGI-S) Score, as Related to Symptoms of Agitation
Description: The severity of agitation for each participant was rated using the CGI-S. The investigator (or designee) answered the following question: "Considering your total clinical experience with this particular population, how mentally ill (as related to agitation) was the participant at the observation period?" Response choices were 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. The score 0 (= not assessed) was set to missing. The CGI-S was therefore a 7-point scale (1-7). The primary analysis used a mixed-effect model repeated measure approach.
Time Frame: From screening to week 12/early termination
Population: The intent-to-treat (ITT) population consisted of all participants in the randomized sample, who took at least 1 dose of the IMP and had a baseline and at least one postbaseline evaluation for the CMAI total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day)
Number analyzed (Participants) | 131 | 135
units on a scale | 4.54 (0.77) | 4.51 (0.74)

ADVERSE EVENTS:
Time Frame: Through the trial: From screening to Week 12 and 30 (+2) days follow-up period.
Description: Only participants who received at least 1 dose of investigational medical product were analyzed for safety (Brexpiprazole N=132).
Arm/Group | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/132 | 1/137
Serious Adverse Events (participants affected / at risk) | 7/132 | 6/137
Other Adverse Events (participants affected / at risk) | 24/132 | 29/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) (N=132) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day) (N=137)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (Flexible Dose Range 0.5 to 2 mg/Day) (N=132) | Placebo (Flexible Dose Range 0.5 to 2 mg/Day) (N=137)
Somnolence (Nervous system disorders) | 8 | 5
Dizziness (Nervous system disorders) | 6 | 7
Headache (Nervous system disorders) | 10 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT01922258/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT01922258/SAP_001.pdf